CLINICAL TRIAL: NCT00433394
Title: Protocol for Registration and Consent to the Childhood Cancer Research Network - A Limited Institution Pilot
Brief Title: Registration and Informed Consent Study for the Childhood Cancer Research Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AADM01P1; COG-AADM01P1 (Other: Children's Oncology Group); NCT00228709 (obsolete NCT alias)
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stratum 1: No Consent for personal identification (Experimental): Data to be collected for this stratum include histology, primary site, treating hospital, and institutional principal investigator. Data will be coded using the North American Association for Central Cancer Registries (N.A.A.C.C.R.) data standards for cancer registries.
  Interventions: Procedure: educational intervention
- Stratum 2: Consent for personal identification - No Contact (Experimental): Data will be collected for this study include:child's name, parent's name, address, telephone number, child's date of birth, race, ethnicity, histology, primary site, treating hospital, and institutional principal investigator. Data will be coded using the North American Association for Central Cancer Registries (N.A.A.C.C.R.) data standards for cancer registries. No contact for future to ask me to consider taking part in Research Network approved studies
  Interventions: Procedure: cancer prevention intervention; Procedure: educational intervention
- Stratum 3: Consent for personal identification - Contact (Experimental): Data will be collected for this study include:child's name, parent's name, address, telephone number, child's date of birth, race, ethnicity, histology, primary site, treating hospital, and institutional principal investigator. Data will be coded using the North American Association for Central Cancer Registries (N.A.A.C.C.R.) data standards for cancer registries Someone from the Childhood Cancer Research Network may contact me in the future to ask me to consider taking part in Research Network approved studies
  Interventions: Procedure: cancer prevention intervention; Procedure: educational intervention

INTERVENTIONS:
Procedure: cancer prevention intervention
  Arms: Stratum 2: Consent for personal identification - No Contact; Stratum 3: Consent for personal identification - Contact
Procedure: educational intervention

SUMMARY:
RATIONALE: Collecting informed consent from parents of children with cancer to register with the Childhood Cancer Research Network may help the study of cancer in the future.

PURPOSE: This study is collecting informed consent to register younger patients with cancer into the Childhood Cancer Research Network.

DETAILED DESCRIPTION:
OBJECTIVES:

* Obtain informed consent from parents (and the child, when appropriate) of children diagnosed with cancer (who are under 21 years of age) to register their child's name and address with the Childhood Cancer Research Network.
* Obtain informed consent from parents (and the child, when appropriate) of children diagnosed with cancer (who are under 21 years of age) to be contacted in the future for possible participation in non-therapeutic research studies involving the parents and/or child.
* Facilitate the systematic registration of pediatric and adolescent patients diagnosed with cancer into the Childhood Cancer Research Network.

OUTLINE: Consent is obtained from parents (and pediatric patients, where applicable) to register the patient's and parent's names and addresses with the Childhood Cancer Research Network, provide a copy of the pathology report to the Network, and contact parents in the future for possible non-therapeutic research studies involving the parents and/or child.

Information provided will be held in strict confidence.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Child (< 21 years of age) with newly diagnosed cancer

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2242 (Actual)
Dates: Start 2001-05; Primary Completion 2007-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Informed consent collection to register with the Childhood Cancer Research Network
Informed consent collection for possible participation in future non-therapeutic research studies
Facilitation of systematic registration into the Childhood Cancer Research Network

CONTACTS AND LOCATIONS:
Overall Officials: Julie A. Ross, PhD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (21):
- United States (19):
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minneapolis, Minneapolis, Minnesota
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Albany Medical Center Hospital, Albany, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec